CLINICAL TRIAL: NCT04822909
Title: A Pilot Study to Evaluate the Efficacy and Safety of Apremilast in Patients of Chronic and Recurrent Erythema Nodosum Leprosum
Brief Title: A Study to Evaluate the Efficacy and Safety of Apremilast in Patients of Chronic and Recurrent Erythema Nodosum Leprosum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Tarun Narang, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK/4917/Study/05
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Erythema Nodosum Leprosum
MeSH Terms: interventions — Tablets; apremilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apremilast group (Experimental): The study patients will be treated with oral apremilast, administered initially a dose of 10 mg once daily, gradually increasing to reach the maximal therapeutic dosage of 30 mg twice daily before end of 1st week of starting the therapy.
  The treatment will be continued till 6 months and we will taper the steroids by 10mg/ 2 weeks till 20mg and then 5 mg/ 2 weeks till discontinuation of steroids.
  Interventions: Drug: Apremilast;Apremilast;Apremilast 10 MG; 20 MG; 30 MG Oral Tablet

INTERVENTIONS:
Drug: Apremilast;Apremilast;Apremilast 10 MG; 20 MG; 30 MG Oral Tablet — The study patients will be treated with oral apremilast, administered initially a dose of 10 mg once daily, gradually increasing to reach the maximal therapeutic dosage of 30 mg twice daily before end of 1st week of starting the therapy.
  The treatment will be continued till 6 months and we will taper the steroids by 10mg/ 2 weeks till 20mg and then 5 mg/ 2 weeks till discontinuation of steroids.
  If a patient worsens after treatment or develops any serious adverse event after initiation of treatment, he will be withdrawn from the study.
  If there is no response to the treatment and we are unable to taper steroids after 12 weeks of therapy then the patient will be withdrawn from the study
  Other Names: Apremilast

SUMMARY:
Leprosy is a chronic infectious disease caused by Mycobacterium leprae. The disease manifests with a varied spectrum, ranging from localized tuberculoid leprosy (TT) to generalized lepromatous leprosy (LL) types. The normal course of leprosy is interrupted by troublesome immune reactions, namely lepra reactions. ENL (a type 2 lepra reaction) is an immune-mediated hypersensitivity reaction, presenting as erythematous, tender, papulo-nodules and associated with constitutional symptoms (fever, arthralgias etc). Pro-inflammatory mediators are elevated, especially tumour necrosis factor α (TNF-α), interferon-γ (IFN- γ) and interleukins (IL-2, IL-6, IL-12). LL type and high bacteriological index are considered to be risk factors for ENL. Lesions usually appear after starting MDT, although it may also be presenting feature. Diagnosis is made by characteristic lesions associated with constitutional symptoms and painful nerve thickening. Mild episodes of ENL respond to adequate rest and oral aspirin. Severe episodes necessitate anti-inflammatory drugs like corticosteroids (e.g. Prednisolone) and/or thalidomide. Use of high-dose prednisolone increases risk of steroid toxicity. Thalidomide is category X drug (unsafe in pregnancy), not freely available and has cost-limitations. Clofazimine requires higher doses, takes 4 to 6 weeks to be effective and produces gastrointestinal side-effects and skin discoloration. Minocycline has been tried as an alternative; however the drug itself has been reported to precipitate ENL in some patients. Thus, a safe and effective steroid-sparing agent for ENL remains elusive.

Cyclic adenosine monophosphate (cAMP) is an intracellular signal molecule. Phosphodiesterases (PDEs) catalyse degradation of cAMP leading to its inactivation. Inhibition of PDEs leads to increased intracellular cAMP, which has anti-inflammatory actions. PDE-4 isoenzymes are the predominant cAMP degrading enzymes in most immune cells. Apremilast is an oral phosphodiesterase-4 (PDE-4) inhibitor currently used clinically for the treatment of psoriasis and other chronic inflammatory diseases. The anti-inflammatory effects of apremilast shown in-vitro includes downregulating TNF-α, IFN-γ, IL-2, IL-12 and IL-23. Although apremilast is not yet clinically indicated in ENL, its anti-inflammatory spectrum targeting the same molecules as those implicated in ENL and efficacy seen in other inflammatory conditions warrants its trial in chronic, recurrent ENL patients.

DETAILED DESCRIPTION:
ENL is confined to leprosy patients classified as BL or LL (Ridley-Jopling), which in turn comprise the multi-bacillary (MB) patient group, as defined by WHO. ENL presents as new, red, painful and tender nodules in the skin, usually on the legs and arms, and sometimes on the trunk. ENL varies in severity. When the reaction is mild, only the skin is affected and there may be low grade fever. When the reaction is severe, the nodules are multiple and may ulcerate, and other organs may be inflamed, such as the nerves, eyes, joints, testes, and lymph nodes. ENL may occur before, during or after MDT treatment, and several years later. It can occur as a single acute episode, but frequently develops into a chronic condition with recurrent episodes. Immune responses causing ENL are triggered by high loads of fragmented bacilli in skin tissue. The complex mechanisms underlying ENL are not fully understood yet which makes treatment difficult.

Treatment of ENL is much debated and a very challenging issue. There is no universally accepted regimen that is fully effective. Most therapies for ENL aim to control the acute inflammation, relieving the pain and preventing further damage or new episodes. Several treatments are available for ENL. The conventional treatment for mild ENL is rest and anti-inflammatory medication. Aspirin was the most commonly used anti-inflammatory medication, but indomethacin, chloroquine and colchicine have been tested as well. There is not much evidence that these drugs are more beneficial than aspirin. For severe ENL, prednisolone, the most widely available corticosteroid, and clofazimine are most commonly used. ENL is often recurrent or chronic and requires high-dose and prolonged courses of prednisolone for disease control. This increases the risk of adverse events, such as hypertension or diabetes, and steroid dependency.

Apremilast is a novel, phosphodiesterase 4 (PDE 4) antagonist, and an orally administered small molecule, acts by specifically targeting a central pathogenic mechanism, binding directly to the PDE-4 enzyme and evading complex antigen-receptor interactive immunoregulatory mechanisms. Apremilast is an immune modulator rather than an immunosuppressant.

Anti-inflammatory actions of Apremilast includes

1. Increased levels of cAMP, which reduces the levels of pro- inflammatory cytokines (such as tumor necrosis factor (TNF)-α, interleukin (IL)-23, IL-12, and leukotriene B4) and also increases the levels of anti-inflammatory cytokines (such as IL-10)
2. Binds to toll-like receptor 4 in peripheral blood mononuclear cells, which further decrease the production of pro-inflammatory cytokines
3. Decreases the activity of nitric oxide synthase Because of its anti-inflammatory actions, Apremilast may have a significant role in the treatment of patients with Erythema Nodosum Leprosum who have not responded to other conventional treatment.

Use and safety of apremilast in other dermatoses Apremilast has been extensively used in dermatology in psoriasis and psoriatic arthropathy and is FDA-approved for both the indications. Multiple randomized controlled trials (RCTs) have shown efficacy of oral apremilast in moderate to severe chronic plaque psoriasis. In an RCT involving 352 adult patients of moderate to severe psoriasis, oral apremilast was well-tolerated, safe and produced significant improvement in psoriasis area and severity index (PASI) scores, when used in dosage of 20 mg twice daily or 30 mg twice daily as compared to placebo and lower doses (p<0.0001).

In another multi-centric RCT in 259 patients of psoriasis, apremilast produced significant reduction in PASI scores over 12 weeks and was well-tolerated20.

In the three programs conducted under the title of Psoriatic Arthritis Long term Assessment of Clinical Efficacy (PALACE), when given in dose of 20 or 30 mg twice daily for 52 weeks, apremilast was significantly effective in improving the swollen joint count and the tender joint counts in psoriatic arthropathy without any serious adverse effects.

In a study performed in 15 patients with cutaneous sarcoidosis, oral apremilast at a dose of 20 mg twice daily, was shown to produce clinical improvement in paired photographs as well as significant decrease in sarcoidosis activity and severity index (SASI) scores with 12 weeks of therapy. The therapy was safe and no serious side-effects were reported.

The most common adverse drug reactions (ADRs) recorded in previous studies were diarrhoea, nausea, upper respiratory tract infection and headache. Other ADRs included dyspepsia, decreased appetite, migraine, back pain, bronchitis etc. However, most of these side effects have a mild to moderate intensity, with a self limiting nature. In a study by Crowley et al, safety findings were reported for 0 to ≥156 weeks from the Efficacy and Safety Trial Evaluating the Effects of Apremilast in Psoriasis (ESTEEM) 1 and 2 and the authors concluded that apremilast had an acceptable safety profile and was well-tolerated despite use for ≥156 weeks. Although there are no reports of use of apremilast in leprosy, the use is not expected to cause any significant adverse effects in view of its relative safe profile in other inflammatory dermatoses.

AIMS AND METHODS

Primary objective To assess the efficacy of apremilast in patients of chronic and recurrent ENL, who have not responded to either clofazimine or minocycline

Secondary objective To evaluate the safety profile and document adverse effects of oral apremilast in chronic recurrent ENL

MATERIALS AND METHODS

Study period: November 2018 to April 2019 Number of patients to be enrolled in pilot study: 10 This will be a pilot study to assess the efficacy and safety of Apremilast in chronic and recurrent Erythema Nodosum Leprosum (ENL) conducted in the department of Dermatology, Venereology and Leprology, PGIMER, Chandigarh after obtaining approval from the institutional ethics committee.

Definitions Erythema Nodosum Leprosum (ENL) is diagnosed when a patient with leprosy has crops of tender subcutaneous skin lesions. Systemic features are recorded separately and include: fever (temperature >38°C), neuritis, joint pain, bone tenderness, orchitis, iritis, oedema, malaise, anorexia and lymphadenopathy

Chronic ENL: ENL occurring for 24 weeks or more during which a patient requires ENL treatment either continuously or where any treatment free period has been 27 days or less.

Recurrent ENL: If a patient experiences a second or subsequent episode of ENL occurring 28 days or more after stopping treatment for ENL

Data collection All the diagnosed patients of chronic and recurrent ENL will be screened for the eligibility. Patients who give consent and fulfil the eligibility criteria in the study period will be consecutively enrolled in the study.

Drug protocol to be used:

Oral tablet of Apremilast 30 mg twice in a day daily for 6 months after an initial titration schedule.

Titration schedule shall be as follows:

The study patients will be treated with oral apremilast, administered initially a dose of 10 mg once daily, gradually increasing to reach the maximal therapeutic dosage of 30 mg twice daily before end of 1st week of starting the therapy.

The treatment will be continued till 6 months and we will taper the steroids by 10mg/ 2 weeks till 20mg and then 5 mg/ 2 weeks till discontinuation of steroids.

If a patient worsens after treatment or develops any serious adverse event after initiation of treatment, he will be withdrawn from the study.

If there is no response to the treatment and we are unable to taper steroids after 12 weeks of therapy then the patient will be withdrawn from the study.

STATISTICAL ANALYSIS The statistical analysis will be carried out using Statistical Package for Social Sciences (SPSS Inc., Chicago, IL, version 20.0 for Windows). All quantitative variables (age, duration of the symptoms, age at onset) will be estimated using measures of central location (mean, median) and measures of dispersion (standard deviation and standard error). Normality of data will be checked by measures of Kolmogorov Smirnov tests of normality. For normally distributed data means will be compared using student's t-test. For skewed data or for scores, Mann-Whitney test will be applied & IQR will also be calculated. For time related variables, Wilcoxon Signed rank test will be applied. Qualitative or categorical variables will be described as frequencies and proportions. Proportions will be compared using Chi square or Fisher's exact test whichever is applicable. All statistical tests will be two-sided and will be performed at a significance level of α=.05.

ETHICAL JUSTIFICATION Apremilast is one of the newer and safe oral therapies currently used for treating patients with severe psoriasis and psoriatic arthropathy due to its anti-inflammatory effects. ENL is an immune-mediated inflammatory response occurring in patients of multibacillary leprosy. Although apremilast targets those inflammatory mediators, which are also implicated in ENL, the exact role and possible efficacy of apremilast in patients with chronic and recurrent ENL is not yet clear and has not been evaluated before. This study aims to study the efficacy and safety of oral apremilast in ENL patients. All patients will be recruited voluntarily after obtaining informed consent. Hence, the study is ethically justified.

Clinical assessment and follow-up visits will be performed during scheduled visits. There will be no financial burden on the patient for the study purpose as apremilast will be provided by the investigators and the patients will not be compensated financially for participating in the study. Treatment of the patient will not be altered by the refusal or agreement of the patient to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic and recurrent ENL cases of leprosy regardless of age, sex and treatment status with MDT
2. Patients not responded with paracetamol, clofazimine, pentoxifylline, colchicine, methotrexate, azathioprine, TNF inhibitors etc.,
3. Patients who can give valid consent.
4. Willing for monthly follow-up visits for at least 3 months.

Exclusion Criteria:

1. Pregnant and lactating mothers
2. Severe renal dysfunction
3. Patients with HIV, Hepatitis B and Hepatitis C
4. Inability to come for monthly follow up visits for 6 months
5. Those who cannot provide consent for the study
6. Known case of psychiatric disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of apremilast in chronic, recurrent erythema nodosum leprosum | 6 months
  Duration taken to attain clinical remission shall be determined in patients with chronic, recurrent erythema nodosum leprosum receiving apremilast

SECONDARY OUTCOMES:
Clinical features of ENL | 6 months
  Clinical characteristics of ENL patients shall be ascertained using ENLIST severity scale
Adverse effects of apremilast | 6 months
  Adverse effects, if any, shall be documented on follow-up in all patients of chronic recurrent erythema nodosum leprosum receiving apremilast

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Narang, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (3):
- India (3):
  - Dermatology OPD, New OPD Building, Level 5C, Postgraduate Institute of Medical Education and Research, Chandigarh
  - PGIMER, Chandigarh
  - Tarun Narang, Chandigarh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parkash O. Classification of leprosy into multibacillary and paucibacillary groups: an analysis. FEMS Immunol Med Microbiol. 2009 Jan;55(1):1-5. doi: 10.1111/j.1574-695X.2008.00491.x. Epub 2008 Nov 13. PMID 19040664
- [Background] Ridley DS, Jopling WH. Classification of leprosy according to immunity. A five-group system. Int J Lepr Other Mycobact Dis. 1966 Jul-Sep;34(3):255-73. No abstract available. PMID 5950347
- [Background] Lockwood DN, Nicholls P, Smith WC, Das L, Barkataki P, van Brakel W, Suneetha S. Comparing the clinical and histological diagnosis of leprosy and leprosy reactions in the INFIR cohort of Indian patients with multibacillary leprosy. PLoS Negl Trop Dis. 2012;6(6):e1702. doi: 10.1371/journal.pntd.0001702. Epub 2012 Jun 26. PMID 22745841
- [Background] Partida-Sanchez S, Favila-Castillo L, Pedraza-Sanchez S, Gomez-Melgar M, Saul A, Estrada-Parra S, Estrada-Garcia I. IgG antibody subclasses, tumor necrosis factor and IFN-gamma levels in patients with type II lepra reaction on thalidomide treatment. Int Arch Allergy Immunol. 1998 May;116(1):60-6. doi: 10.1159/000023926. PMID 9623511
- [Background] Van Veen NH, Lockwood DN, van Brakel WH, Ramirez J Jr, Richardus JH. Interventions for erythema nodosum leprosum. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD006949. doi: 10.1002/14651858.CD006949.pub2. PMID 19588412
- [Background] Schafer PH, Parton A, Gandhi AK, Capone L, Adams M, Wu L, Bartlett JB, Loveland MA, Gilhar A, Cheung YF, Baillie GS, Houslay MD, Man HW, Muller GW, Stirling DI. Apremilast, a cAMP phosphodiesterase-4 inhibitor, demonstrates anti-inflammatory activity in vitro and in a model of psoriasis. Br J Pharmacol. 2010 Feb;159(4):842-55. doi: 10.1111/j.1476-5381.2009.00559.x. Epub 2009 Dec 24. PMID 20050849
- [Background] Papp K, Cather JC, Rosoph L, Sofen H, Langley RG, Matheson RT, Hu C, Day RM. Efficacy of apremilast in the treatment of moderate to severe psoriasis: a randomised controlled trial. Lancet. 2012 Aug 25;380(9843):738-46. doi: 10.1016/S0140-6736(12)60642-4. Epub 2012 Jun 29. PMID 22748702
- [Background] Kavanaugh A, Mease PJ, Gomez-Reino JJ, Adebajo AO, Wollenhaupt J, Gladman DD, Hochfeld M, Teng LL, Schett G, Lespessailles E, Hall S. Longterm (52-week) results of a phase III randomized, controlled trial of apremilast in patients with psoriatic arthritis. J Rheumatol. 2015 Mar;42(3):479-88. doi: 10.3899/jrheum.140647. Epub 2015 Jan 15. PMID 25593233
- [Background] Crowley J, Thaci D, Joly P, Peris K, Papp KA, Goncalves J, Day RM, Chen R, Shah K, Ferrandiz C, Cather JC. Long-term safety and tolerability of apremilast in patients with psoriasis: Pooled safety analysis for >/=156 weeks from 2 phase 3, randomized, controlled trials (ESTEEM 1 and 2). J Am Acad Dermatol. 2017 Aug;77(2):310-317.e1. doi: 10.1016/j.jaad.2017.01.052. Epub 2017 Apr 14. PMID 28416342
- [Background] Walker SL, Sales AM, Butlin CR, Shah M, Maghanoy A, Lambert SM, Darlong J, Rozario BJ, Pai VV, Balagon M, Doni SN, Hagge DA, Nery JAC, Neupane KD, Baral S, Sangma BA, Alembo DT, Yetaye AM, Hassan BA, Shelemo MB, Nicholls PG, Lockwood DNJ; Erythema Nodosum Leprosum International STudy Group. A leprosy clinical severity scale for erythema nodosum leprosum: An international, multicentre validation study of the ENLIST ENL Severity Scale. PLoS Negl Trop Dis. 2017 Jul 3;11(7):e0005716. doi: 10.1371/journal.pntd.0005716. eCollection 2017 Jul. PMID 28671966